CLINICAL TRIAL: NCT06682585
Title: Determination of Nutritional Status of Duchenne Muscular Dystrophy Patients and Evaluation of the Effectiveness of Disease-Specific Nutrition Therapy
Brief Title: Nutritional Status and Therapy in DMD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Betül ULU, Principal Investigator, Dietitian, PhD Student, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 111-659-22
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-11

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Duchenne Muscular Dystrophy; Nutrition
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Intervention (Experimental): The participants of the arm will follow diet program specially prepared for them for 12 weeks.
  Interventions: Other: Individualised dietary intervention

INTERVENTIONS:
Other: Individualised dietary intervention — * Energy Intake: Caloric needs will be calculated based on the patient's age, weight, and activity level, taking into account the potential impact of corticosteroid therapy on energy expenditure.
  * Protein Intake: Protein requirements will be met through a balanced diet, aiming to optimize muscle protein synthesis.
  * Calcium and Vitamin D Intake: Adequate intake of these nutrients will be emphasized to support bone health and prevent osteoporosis.
  * Fluid Intake: Fluid intake will be monitored to prevent dehydration and constipation.
  * Carbohydrate Intake: A low-glycemic index diet will be recommended to manage blood glucose levels and insulin resistance, especially in patients on corticosteroid therapy.
  * Sodium Intake: Sodium intake will be restricted to minimize fluid retention and hypertension.

SUMMARY:
Brief Summary

The goal of this clinical trial is to evaluate the impact of a disease-specific, individualized diet on the nutritional status and functional abilities of Duchenne muscular dystrophy (DMD) patients. The study will focus on children aged 4-8 years residing in Ankara, Turkey.

Key questions the investigators aim to answer:

Can a tailored dietary intervention improve the nutritional status of DMD patients? Does a specialized diet positively impact the functional abilities of DMD patients, as measured by the North Star Ambulation Assessment (NSAA)? Participants will undergo a comprehensive nutritional assessment, including anthropometric measurements, and will receive individualized dietary counseling. The intervention will focus on optimizing energy, protein, calcium, and fluid intake, as well as addressing the potential side effects of corticosteroid therapy.

The primary outcome measure will be changes in nutritional status, as assessed by anthropometric measurements. Secondary outcome measures will include changes in functional abilities as measured by the NSAA and quality of life assessments.

DETAILED DESCRIPTION:
Study Objective This study aims to investigate the efficacy of a disease-specific, individualized dietary intervention in improving the nutritional status and functional abilities of Duchenne Muscular Dystrophy (DMD) patients aged 4-8 years residing in Ankara, Turkey.

Study Design This is a prospective, interventional study. Intervention

A 12-week individualized dietary intervention will be implemented for each participant. The intervention will focus on:

* Energy Intake: Caloric needs will be calculated based on the patient's age, weight, and activity level, taking into account the potential impact of corticosteroid therapy on energy expenditure.
* Protein Intake: Protein requirements will be met through a balanced diet, aiming to optimize muscle protein synthesis.
* Calcium and Vitamin D Intake: Adequate intake of these nutrients will be emphasized to support bone health and prevent osteoporosis.
* Fluid Intake: Fluid intake will be monitored to prevent dehydration and constipation.
* Carbohydrate Intake: A low-glycemic index diet will be recommended to manage blood glucose levels and insulin resistance, especially in patients on corticosteroid therapy.
* Sodium Intake: Sodium intake will be restricted to minimize fluid retention and hypertension.

Outcome Measures Changes in anthropometric measurements (body weight, height, BMI, skinfold measurements) Changes in functional abilities as assessed by the North Star Ambulation Assessment (NSAA) Changes in functional abilities as assessed by handgrip strenght Changes in micro and micro nutrient intake as assessed by three-day food consumption record Data Collection Data will be collected through face-to-face interviews with parents or primary caregivers and patients with DMD. After the first interview, a second interview will be conducted 12 weeks after the personalized diet has been planned.

Baseline Assessment:

* Demographic information
* Medical history
* Nutritional assessment (anthropometric measurements, dietary intake assessment)
* Functional assessment (NSAA)

Follow-up Assessments:

* Anthropometric measurements
* Functional assessment (NSAA)
* Dietary intake assessment Data Analysis Statistical analysis will be performed using appropriate statistical software. Descriptive statistics will be used to summarize the baseline characteristics of the participants. Parametric or non-parametric tests will be used to compare pre- and post-intervention outcomes, as appropriate.

Ethical Considerations The study will be conducted in accordance with the Declaration of Helsinki and approved by the local ethics committee. Informed consent will be obtained from the parents or legal guardians of the participants.

By addressing the specific nutritional needs of DMD patients, this study aims to improve their overall health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Duchenne Muscular Dystrophy (DMD) Must be between 4 and 8 years old Able to ambulate independently Must be residing in Ankara province, Turkey Must be willing to participate and adhere to the dietary intervention, as confirmed by both the patient and their legal guardian(s) Must be currently receiving corticosteroid therapy

Exclusion Criteria:

Inability to read and write in Turkish Wheelchair-bound or unable to ambulate independently Significant liver or kidney dysfunction Scheduled for major surgery within 6 months of study enrollment Symptoms of dysphagia and swallowing difficulties Significant respiratory distress or respiratory insufficiency requiring mechanical ventilation.

Ages: 48 Months to 96 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Duchenne Muscular Dystrophy is caused by a defect in the dystrophin gene encoded in the Xp21 region of the X chromosome. Since it originates from the X chromosome, it is inherited from the mother, and while boys develop the disease, girls continue their lives as carriers.
Enrollment: 9 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements | From enrollment to the end of diet at 12 weeks
  Changes in body weight (kg). Body weight will be measured with an electronic scale sensitive to 0.1 kilograms.
Anthropometric measurements | From enrollment to the end of diet at 12 weeks
  Changes in skinfold thickness (triceps, biceps, subscapular, and suprailiac) (in millimeters) Skinfold thickness will be compared to the World Health Organization's percentile and Z score charts to determine adequacy, deficiency, or excess.
Anthropometric measurements | From enrollment to the end of diet at 12 weeks
  Changes in height (cm). Height is measured with the individual standing upright and the head in the Frankfurt plane (the orbitale point and tragion point are set to be on the horizontal plane), while the vertical distance from the ground to the vertex, which is the highest point of the head, will be measured with a tape measure on a fixed plane.
Anthropometric measurements | From enrollment to the end of diet at 12 weeks
  Changes in Body Mass Index (BMI)(kg/m²). BMI will be obtained by dividing the particioant's body weight in kg by the square of the height in meters.
  Body mass index will be evaluated with the World Health Organization's percentile and Z score charts.

SECONDARY OUTCOMES:
Functional Ability | From enrollment to the end of diet at 12 weeks
  Changes in the North Star Ambulation Assessment (NSAA) score meausered by a specialist physiotherapist. The total score varies between 0-34. A higher score indicates better ambulation and motor function.
Functional Ability | From enrollment to the end of diet at 12 weeks
  Changes in hand grip strength measured by hand dynamometry (in kilograms)

OTHER OUTCOMES:
Dietary Adherence | From enrollment to the end of diet at 12 weeks
  After the dietary intervention, 3-day food consumption records will be taken again. The 3-day food consumption records before and after the dietary intervention will be examined. The compatibility of the latest consumption records with the macro and micronutrients of the recommended diet and the differences between the first 3-day food consumption record will be examined. The computer program called BeBIS will be used for the analysis of macro and micronutrients.

CONTACTS AND LOCATIONS:
Locations (1):
- DMD Aileleri Derneği, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Summer SS, Wong BL, Rutter MM, Horn PS, Tian C, Rybalsky I, Shellenbarger KC, Kalkwarf HJ. Age-related changes in appendicular lean mass in males with Duchenne muscular dystrophy: A retrospective review. Muscle Nerve. 2021 Feb;63(2):231-238. doi: 10.1002/mus.27107. Epub 2020 Dec 7. PMID 33104257
- [Background] Guzikowska E, Markiewicz-Loskot G, Hercog R. [Serum opsonization activity in children with recurrent respiratory tract infections]. Pediatr Pol. 1986 Dec;61(12):780-3. No abstract available. Polish. PMID 3601481
- [Background] Billich N, Evans M, Truby H, Ryan MM, Davidson ZE. The association between dietary factors and body weight and composition in boys with Duchenne muscular dystrophy. J Hum Nutr Diet. 2022 Oct;35(5):804-815. doi: 10.1111/jhn.12987. Epub 2022 Feb 1. PMID 34936149
- [Background] de Souza Costa AD, Vermeulen-Serpa KM, Batista Marinho KM, Carvalho Xavier de Medeiros CA, Antunes de Araujo A, Teixeira Dourado-Junior ME, Brandao-Neto J, Lima Maciel BL, Helena de Lima Vale S. Persistent inflammation and nutritional status in Duchenne muscular dystrophy. Clin Nutr ESPEN. 2024 Jun;61:393-398. doi: 10.1016/j.clnesp.2024.04.014. Epub 2024 Apr 20. PMID 38777460
- [Background] Chou E, Lindeback R, D'Silva AM, Sampaio H, Neville K, Farrar MA. Growth and nutrition in pediatric neuromuscular disorders. Clin Nutr. 2021 Jun;40(6):4341-4348. doi: 10.1016/j.clnu.2021.01.013. Epub 2021 Jan 22. PMID 33551221
- [Background] Davidson ZE, Ryan MM, Kornberg AJ, Sinclair K, Cairns A, Walker KZ, Truby H. Observations of body mass index in Duchenne muscular dystrophy: a longitudinal study. Eur J Clin Nutr. 2014 Aug;68(8):892-7. doi: 10.1038/ejcn.2014.93. Epub 2014 May 14. PMID 24824013
- [Background] Duan D, Goemans N, Takeda S, Mercuri E, Aartsma-Rus A. Duchenne muscular dystrophy. Nat Rev Dis Primers. 2021 Feb 18;7(1):13. doi: 10.1038/s41572-021-00248-3. PMID 33602943
- [Background] Garcia-Rodriguez R, Hiller M, Jimenez-Gracia L, van der Pal Z, Balog J, Adamzek K, Aartsma-Rus A, Spitali P. Premature termination codons in the DMD gene cause reduced local mRNA synthesis. Proc Natl Acad Sci U S A. 2020 Jul 14;117(28):16456-16464. doi: 10.1073/pnas.1910456117. Epub 2020 Jul 2. PMID 32616572
- [Background] Aartsma-Rus A, Van Deutekom JC, Fokkema IF, Van Ommen GJ, Den Dunnen JT. Entries in the Leiden Duchenne muscular dystrophy mutation database: an overview of mutation types and paradoxical cases that confirm the reading-frame rule. Muscle Nerve. 2006 Aug;34(2):135-44. doi: 10.1002/mus.20586. PMID 16770791
- [Background] Mercuri E, Bonnemann CG, Muntoni F. Muscular dystrophies. Lancet. 2019 Nov 30;394(10213):2025-2038. doi: 10.1016/S0140-6736(19)32910-1. PMID 31789220
- [Background] Davis J, Samuels E, Mullins L. Nutrition Considerations in Duchenne Muscular Dystrophy. Nutr Clin Pract. 2015 Aug;30(4):511-21. doi: 10.1177/0884533615586202. Epub 2015 May 14. PMID 25977513
- [Background] Bernabe-Garcia M, Rodriguez-Cruz M, Atilano S, Cruz-Guzman ODR, Almeida-Becerril T, Calder PC, Gonzalez J. Body composition and body mass index in Duchenne muscular dystrophy: Role of dietary intake. Muscle Nerve. 2019 Mar;59(3):295-302. doi: 10.1002/mus.26340. Epub 2018 Dec 12. PMID 30194761